CLINICAL TRIAL: NCT00810264
Title: CELESTIAL Post Approval Registry: Corox OTW, Endocardial, Left Ventricular Steroid Lead, Bipolar Post Approval Registry
Brief Title: Post Approval Registry of Corox OTW, Endocardial, Left Ventricular Steroid Lead, Bipolar
Acronym: CELESTIAL
Status: Completed | Type: Observational
Sponsor: Biotronik, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CELESTIAL
Record Dates: First submitted 2008-12-17; First posted 2008-12-18 (Estimated); Results first posted 2019-11-29 (Actual); Last update posted 2019-11-29 (Actual); Status verified 2019-11

CONDITIONS: Congestive Heart Failure
Keywords: Long-term safety and reliability of a bipolar left ventricular lead on congestive heart failure patients
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Data Collection Group
  Interventions: Device: CRT Therapy - LV Lead Registry

INTERVENTIONS:
Device: CRT Therapy - LV Lead Registry — Collecting long-term safety and efficacy data on a market-released left ventricular lead.

SUMMARY:
The objective of this study is to confirm the long-term safety and reliability of the Corox OTW BP left ventricular (LV) pacing lead. As a condition of approval, the FDA required that a registry documenting the post approval clinical experience of these leads be designed and implemented.

DETAILED DESCRIPTION:
This study is an FDA-required, multi-center, prospective, non-randomized, data collection registry. Eligible patients must have been successfully implanted with a Corox OTW BP, Corox OTW-S BP, or Corox OTW-L BP LV lead with a BIOTRONIK CRT device and consented and enrolled between 7-180 days following implant. At least 2500 patients will be enrolled in this post-approval registry, and each patient will be followed for five years post-implant.

Safety will be evaluated based on the analysis of the overall incidence of lead-related adverse events that require additional invasive intervention. In addition, each individual adverse event will be separately investigated. Lead parameters for sensing, pacing thresholds, and impedance will also be evaluated. Reporting of all adverse events will be performed twice a year in order to identify and characterize any trends in adverse events, failure modes, or failure rates.

ELIGIBILITY:
Inclusion Criteria:

* Successfully implanted BIOTRONIK CRT system, including a Corox BP LV lead, from 7-180 days prior to enrollment
* Able to understand the nature of the registry and give informed consent
* Available for follow-up visits on a regular basis at the investigational site
* Age greater than or equal to 18 years

Exclusion Criteria:

* Enrolled in any IDE clinical study
* Planned cardiac surgical procedures or interventional measures within the next 6 months
* Expected to receive a heart transplant within 1 year
* Life expectancy less than 1 year
* Presence of another life-threatening, underlying illness separate from their cardiac disorder
* Pregnancy
* Inability to provide date of implant, devices implanted, age, gender, and whether the patient experienced any protocol-defined adverse events since implant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be obtained from the investigators' general patient population according to the inclusion and exclusion criteria described below.
Sampling Method: Non-Probability Sample
Enrollment: 2499 (Actual)
Dates: Start 2008-12; Primary Completion 2018-11-02 (Actual); Study Completion 2018-11-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (86):
- United States (86):
  - Birmingham, Alabama
  - Glendale, Arizona
  - Mesa, Arizona
  - Phoenix, Arizona
  - Scottsdale, Arizona
  - Tucson, Arizona
  - Anaheim, California
  - Fairfield, California
  - Fountain Valley, California
  - Glendale, California
  - Hawthorne, California
  - Inglewood, California
  - Los Angeles, California
  - National City, California
  - Northridge, California
  - Orange, California
  - Rancho Mirage, California
  - Santa Barbara, California
  - Torrance, California
  - Ventura, California
  - Watsonville, California
  - Aurora, Colorado
  - Boulder, Colorado
  - Danbury, Connecticut
  - Brooksville, Florida
  - Davenport, Florida
  - Melbourne, Florida
  - Naples, Florida
  - New Smyrna Beach, Florida
  - St. Petersburg, Florida
  - Tampa, Florida
  - Macon, Georgia
  - Urbana, Illinois
  - Fort Wayne, Indiana
  - Valparaiso, Indiana
  - Owensboro, Kentucky
  - Covington, Louisiana
  - Hammond, Louisiana
  - Lafayette, Louisiana
  - Bangor, Maine
  - Baltimore, Maryland
  - Cumberland, Maryland
  - Lanham, Maryland
  - Rockville, Maryland
  - Burlington, Massachusetts
  - Worcester, Massachusetts
  - Ann Arbor, Michigan
  - Lansing, Michigan
  - Lapeer, Michigan
  - Saginaw, Michigan
  - Wyoming, Michigan
  - Ypsilanti, Michigan
  - Tupelo, Mississippi
  - Crystal City, Missouri
  - St Louis, Missouri
  - Las Vegas, Nevada
  - Glen Ridge, New Jersey
  - New York, New York
  - Rochester, New York
  - Gastonia, North Carolina
  - Winston-Salem, North Carolina
  - Columbus, Ohio
  - Middletown, Ohio
  - Steubenville, Ohio
  - Toledo, Ohio
  - Oklahoma City, Oklahoma
  - Salem, Oregon
  - Chinchilla, Pennsylvania
  - Lancaster, Pennsylvania
  - Philadelphia, Pennsylvania
  - Pottstown, Pennsylvania
  - Yardley, Pennsylvania
  - Columbia, South Carolina
  - Greenville, South Carolina
  - Spartanburg, South Carolina
  - Chattanooga, Tennessee
  - Amarillo, Texas
  - Brownsville, Texas
  - Corpus Christi, Texas
  - Dallas, Texas
  - Kingwood, Texas
  - McKinney, Texas
  - Nacogdoches, Texas
  - Fredericksburg, Virginia
  - Spokane, Washington
  - Yakima, Washington

REFERENCES:
- [Derived] Good ED, Cakulev I, Orlov MV, Hirsh D, Simeles J, Mohr K, Moll P, Bloom H. Long-Term Evaluation of Biotronik Linox and Linox(smart) Implantable Cardioverter Defibrillator Leads. J Cardiovasc Electrophysiol. 2016 Jun;27(6):735-42. doi: 10.1111/jce.12971. Epub 2016 May 3. PMID 26990515

RESULTS

PARTICIPANT FLOW:
Groups:
- BIOTRONIK Corox BP LV Lead: Subjects consented and implanted with a BIOTRONIK Corox BP LV lead.
Period: Overall Study
Arm/Group | BIOTRONIK Corox BP LV Lead
Started | 2499
Completed | 946
Not Completed | 1553
Not completed — Lost to Follow-up | 191
Not completed — Withdrawal by subject or physician | 721
Not completed — Death | 641

BASELINE CHARACTERISTICS:
Population: Baseline characteristics are provided when available, subjects without available baseline characteristics are not included in the number of participants analyzed in this section.
Arm/Group | BIOTRONIK Corox BP LV Lead
Number analyzed (Participants) | 2498
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.4 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 724
  Male | 1774
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 1805
  Hispanic or Latino | 244
  Black or African American | 220
  Asian | 36
  Native Hawaiian or Other Pacific Islander | 7
  American Indian or Alaska Native | 4
  Unknown | 65
  Not Reported | 117
Height [Mean (Standard Deviation); unit: inches] | 67.7 (4.2)
Weight [Mean (Standard Deviation); unit: pounds] | 194.4 (48.1)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects Who Are Free of Complications Related to the Corox LV Lead
Description: The overall incidence of serious adverse events that require additional invasive intervention to resolve, related to the Corox BP LV leads implanted with either BIOTRONIK CRT-P or CRT-D devices.This was evaluated as a serious adverse event free-rate (SAEFR).
Time Frame: 5 years
Population: The evaluable subject population is the sum of the total unique subjects who completed the 5-year follow-up and/or who experienced a primary endpoint adverse event.
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | BIOTRONIK Corox BP LV Lead
Number analyzed (Participants) | 946
percentage of subjects | 94.19 [92.50 to 95.59]
Statistical Analysis 1: Comparison: BIOTRONIK Corox BP LV Lead; Test type: Non-Inferiority — The primary safety endpoint 1 hypothesis was evaluated by performing an exact, non-inferiority test comparing a binomial proportion (overall SAEFR at 5 years) to 92.5%, with a non-inferiority delta of 5%; p < 0.0001, Binomial Proportion

2. Primary Outcome: Percentage of Subjects Experiencing Individual Complications
Description: Evaluation of the individual types of serious adverse events contributing to primary outcome 1.
Time Frame: 5 years
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | BIOTRONIK Corox BP LV Lead
Number analyzed (Participants) | 946
percentage of subjects
  Lead dislodgement (>180 days post-implant) | 3.28 [2.24 to 4.62]
  Abnormal pacing impedance | 1.90 [1.13 to 2.99]
  Conductor fracture | 0.53 [0.17 to 1.23]
  Malposition, excess slack | 0.11 [0.00 to 0.59]

3. Secondary Outcome: Mean Successful Biventricular Pacing in Subjects at the 5 Year In-office Visit.
Description: Successful biventricular pacing in a BIOTRONIK CRT device at scheduled CELESTIAL registry follow-up visits through 5 years post-implant.
Time Frame: 5 years
Population: The subjects analyzed in this outcome must have been consented, implanted with a BIOTRONIK Corox BP LV lead, and completed an in-office 5 year visit. Subjects who did not complete an in-office 5 year visit are excluded from this analysis population.
Measure: Mean (Standard Deviation); unit: percentage of CRT pacing
Groups:
- BIOTRONIK Corox BP LV Lead: Subjects consented and implanted with a BIOTRONIK Corox BP LV lead completing an in-office 5 year visit.
Arm/Group | BIOTRONIK Corox BP LV Lead
Number analyzed (Participants) | 611
percentage of CRT pacing | 97.4 (8.4)

4. Secondary Outcome: Percentage of Subjects Experiencing Serious Adverse Event Excluded From Primary Safety Endpoint
Description: Serious adverse event rates for SAEs excluded from primary safety endpoint through 5 years post-implant.
Time Frame: 5 years
Measure: Number; unit: Percent of subjects
Arm/Group | BIOTRONIK Corox BP LV Lead
Number analyzed (Participants) | 2499
Percent of subjects
  LV lead cardiac perforation | 0.04
  LV lead high pacing threshold, no lead capture | 0.96
  LV lead diaphragmatic / pectoral stimulation | 1.00
  LV lead dislodgement (<180 days post-implant) | 1.64
  RV pacing lead related adverse event | 0.16
  Device related adverse event | 0.28
  Other adverse event | 1.36
  RA lead related adverse event | 2.08
  Implant procedure related adverse event | 3.20
  ICD lead related adverse event | 3.96
  Other high pacing threshold | 0.04

5. Secondary Outcome: Corox BP LV Lead Pacing Threshold Measurements
Description: Pacing threshold measurements for the all Corox BP LV lead models at scheduled CELESTIAL registry through 5 years post-implant.
Time Frame: 5 years
Measure: Mean (Standard Deviation); unit: V
Arm/Group | BIOTRONIK Corox BP LV Lead
Number analyzed (Participants) | 2499
V | 1.41 (1.09)

6. Secondary Outcome: Corox BP LV Lead Sensing Measurements
Description: Sensing measurements for the all Corox BP LV lead models at scheduled CELESTIAL registry through 5 years post-implant.
Time Frame: 5 years
Measure: Mean (Standard Deviation); unit: mV
Arm/Group | BIOTRONIK Corox BP LV Lead
Number analyzed (Participants) | 2499
mV | 13.94 (7.51)

7. Secondary Outcome: Corox BP LV Lead Impedance Measurements
Description: Impedance measurements for the all Corox BP LV lead models at scheduled CELESTIAL registry through 5 years post-implant.
Time Frame: 5 years
Measure: Mean (Standard Deviation); unit: ohms
Arm/Group | BIOTRONIK Corox BP LV Lead
Number analyzed (Participants) | 2499
ohms | 726.5 (250.9)

8. Secondary Outcome: Pacing Threshold Measurements Per Corox BP LV Lead Model
Description: Pacing threshold measurements for the Corox OTW BP LV lead, the Corox OTW-S BP LV lead, and the Corox OTW-L BP LV lead.
Time Frame: 5 years
Measure: Mean (Standard Deviation); unit: V
Groups:
- Corox OTW BP: Subjects consented and originally implanted with a Corox OTW BP lead.
- Corox OTW-S BP: Subjects consented and originally implanted with a Corox OTW-S BP lead.
- Corox OTW-L BP: Subjects consented and originally implanted with a Corox OTW-L BP lead.
Arm/Group | Corox OTW BP | Corox OTW-S BP | Corox OTW-L BP
Number analyzed (Participants) | 686 | 1129 | 684
V | 1.30 (1.01) | 1.40 (1.09) | 1.53 (1.17)

9. Secondary Outcome: Sensing Measurements Per Corox BP LV Lead Model
Description: Sensing measurements for the Corox OTW BP LV lead, the Corox OTW-S BP LV lead, and the Corox OTW-L BP LV lead.
Time Frame: 5 years
Measure: Mean (Standard Deviation); unit: mV
Arm/Group | Corox OTW BP | Corox OTW-S BP | Corox OTW-L BP
Number analyzed (Participants) | 686 | 1129 | 684
mV | 14.82 (7.74) | 13.94 (7.59) | 13.04 (7.02)

10. Secondary Outcome: Impedance Measurements Per Corox BP LV Lead Model
Description: Impedance measurements for the Corox OTW BP LV lead, the Corox OTW-S BP LV lead, and the Corox OTW-L BP LV lead.
Time Frame: 5 years
Measure: Mean (Standard Deviation); unit: ohms
Arm/Group | Corox OTW BP | Corox OTW-S BP | Corox OTW-L BP
Number analyzed (Participants) | 686 | 1129 | 684
ohms | 730.3 (264.9) | 734.4 (251.7) | 709.2 (233.1)

11. Secondary Outcome: Overall Incidence of Primary Endpoint 1 Serious Adverse Events for Each Corox BP Lead Model
Description: Overall incidence of serious adverse events that meet the primary endpoint 1 criteria will be evaluated separately for each Corox BP lead model.
Time Frame: 5 years
Population: The evaluable subject population for each group is the sum of the total unique subjects who completed the 5-year follow-up and/or who experienced a primary endpoint adverse event in the group.
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Corox OTW BP | Corox OTW-S BP | Corox OTW-L BP
Number analyzed (Participants) | 279 | 401 | 266
percentage of subjects | 7.17 [4.43 to 10.85] | 6.48 [4.28 to 9.36] | 3.38 [1.56 to 6.33]

12. Secondary Outcome: Incidence of Individual Types of Primary Endpoint 2 Adverse Events Will be Evaluated Separately for Each Corox BP Lead Model
Description: Incidence of individual types of serious adverse events contributing to primary endpoint 2 will be evaluated separately for each Corox BP lead model.
Time Frame: 5 years
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Corox OTW BP | Corox OTW-S BP | Corox OTW-L BP
Number analyzed (Participants) | 279 | 401 | 266
percentage of subjects
  Lead dislodgement (>180 days post-implant) | 3.58 [1.73 to 6.49] | 3.49 [1.92 to 5.79] | 2.63 [1.06 to 5.35]
  Abnormal pacing impedance | 1.79 [0.58 to 4.13] | 2.99 [1.56 to 5.17] | 0.38 [0.01 to 2.08]
  Conductor fracture | 1.79 [0.58 to 4.13] | 0 [NA to NA] — Unable to obtain confidence interval for 0 subjects | 0 [NA to NA] — Unable to obtain confidence interval for 0 subjects
  Malposition, excess slack | 0 [NA to NA] — Unable to obtain confidence interval for 0 subjects | 0 [NA to NA] — Unable to obtain confidence interval for 0 subjects | 0.38 [0.01 to 2.08]

ADVERSE EVENTS:
Time Frame: Implant to study exit (up to 5 years post-implant)
Arm/Group | BIOTRONIK Corox BP LV Lead
All-Cause Mortality (participants affected / at risk) | 641/2499
Serious Adverse Events (participants affected / at risk) | 281/2499
Other Adverse Events (participants affected / at risk) | 83/2499
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BIOTRONIK Corox BP LV Lead (N=2499)
CHF (Cardiac disorders) | 1 (1)
Device migration (Cardiac disorders) | 2 (2)
Hypotensive arrest / hemodynamic collapse (Cardiac disorders) | 1 (1)
ICD lead T-wave oversensing (Cardiac disorders) | 1 (1)
ICD lead cardiac perforation with or without tamponade (Cardiac disorders) | 1 (1)
ICD lead dislodgement (Cardiac disorders) | 34 (34)
ICD lead high pacing threshold, intermittent capture, no lead capture (Cardiac disorders) | 14 (14)
ICD lead impedance out of range, high impedance, potential conductor fracture (Cardiac disorders) | 15 (15)
ICD lead impedance out of range, low Impedance, potential insulation break (Cardiac disorders) | 11 (11)
ICD lead inability to defibrillate or pace (Cardiac disorders) | 1 (1)
ICD lead oversensing or lead noise (Cardiac disorders) | 10 (10)
ICD lead undersensing or loss of sensing (Cardiac disorders) | 1 (1)
ICD lead, Riata lead externalized (Cardiac disorders) | 2 (2)
ICD lead, unknown, inadequate source documentation (Cardiac disorders) | 1 (1)
Inappropriate shocks (Cardiac disorders) | 1 (1)
LV lead abnormal pacing impedance, high impedance (Cardiac disorders) | 12 (12)
LV lead cardiac perforation with or without tamponade (Cardiac disorders) | 1 (1)
LV lead conductor fracture (Cardiac disorders) | 5 (5)
LV lead dislodgement (Cardiac disorders) | 61 (65)
LV lead excess slack (Cardiac disorders) | 1 (1)
LV lead high pacing threshold, intermittent capture, no lead capture (Cardiac disorders) | 14 (14)
LV lead related diaphgramatic / pectoral stimulation (Cardiac disorders) | 14 (14)
Non-functioning RA lead (Cardiac disorders) | 1 (1)
Pocket pain (Cardiac disorders) | 1 (1)
RA lead dislodgement (Cardiac disorders) | 29 (30)
RA lead high pacing threshold, intermittent capture, no lead capture (Cardiac disorders) | 3 (3)
RA lead impedance out of range, high impedance, potential conductor fracture (Cardiac disorders) | 8 (8)
RA lead impedance out of range, low impedance, potential insulation break (Cardiac disorders) | 1 (1)
RA lead oversensing or lead noise (Cardiac disorders) | 1 (1)
RA lead undersensing or loss of sensing (Cardiac disorders) | 2 (2)
RV pacing lead dislodgement (Cardiac disorders) | 2 (2)
RV pacing lead impedance out of range, high impedance, potential conductor fracture (Cardiac disorders) | 1 (1)
RV pacing lead noise (Cardiac disorders) | 1 (1)
Suspected generator failure requiring opening of pulse generator pocket (Cardiac disorders) | 1 (1)
Twiddler's syndrome (General disorders) | 7 (9)
Implant procedure related infection (Infections and infestations) | 19 (19)
Pocket infection (Infections and infestations) | 2 (2)
Secondary infection (Infections and infestations) | 15 (15)
Skin erosion (Skin and subcutaneous tissue disorders) | 3 (3)
Trauma related dehiscence (Skin and subcutaneous tissue disorders) | 2 (2)
Cardiac perforation with or without tamponade (Surgical and medical procedures) | 1 (1)
Hematoma (Surgical and medical procedures) | 15 (15)
High defibrillation thresholds due to inappropriate lead placement (Surgical and medical procedures) | 1 (1)
Implant procedure related damage to the lead (Surgical and medical procedures) | 1 (1)
LV lead dislodgement during RV lead extraction (Surgical and medical procedures) | 1 (1)
Loose set screw (Surgical and medical procedures) | 5 (5)
Non-healing pocket dehiscence requiring intervention (Surgical and medical procedures) | 8 (8)
Open heart surgery causing LV lead dislodgement (Surgical and medical procedures) | 1 (1)
Persistent arm of unknown cause (Surgical and medical procedures) | 1 (1)
Pneumothorax (Surgical and medical procedures) | 2 (2)
Pocket pain (Surgical and medical procedures) | 2 (2)
RA lead dislodgement during LV lead placement (Surgical and medical procedures) | 1 (1)
SVC perforation during laser lead extraction (Surgical and medical procedures) | 1 (1)
Subclavian vein occlusion (Surgical and medical procedures) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BIOTRONIK Corox BP LV Lead (N=2499)
Arrhythmias (Surgical and medical procedures) | 1 (1)
Coronary sinus dissection (Surgical and medical procedures) | 3 (3)
Diaphragmatic stimulation (Surgical and medical procedures) | 1 (1)
Hematoma (Surgical and medical procedures) | 22 (22)
ICD lead high pacing threshold, intermittent capture, no lead capture (Cardiac disorders) | 2 (2)
ICD lead oversensing (Cardiac disorders) | 2 (2)
ICD lead oversensing or lead noise (Cardiac disorders) | 4 (4)
Incompletely healed incision (Surgical and medical procedures) | 1 (1)
LV lead abnormal pacing impedance, high impedance (Cardiac disorders) | 7 (7)
LV lead dislodgement (Cardiac disorders) | 9 (9)
High pacing threshold (Cardiac disorders) | 1 (1)
LV lead high pacing threshold, intermittent capture, no lead capture (Cardiac disorders) | 10 (10)
LV lead related diaphgramatic / pectoral stimulation (Cardiac disorders) | 11 (11)
Left subclavian vein thrombosis (Surgical and medical procedures) | 1 (1)
Non-healing pocket dehiscence requiring intervention (Surgical and medical procedures) | 1 (1)
RA lead dislodgement (Cardiac disorders) | 1 (1)
RA lead high pacing threshold, intermittent capture, no lead capture (Cardiac disorders) | 3 (3)
RA lead impedance out of range, high impedance, potential conductor fracture (Cardiac disorders) | 1 (1)
RA lead impedance out of range, low impedance, potential insulation break (Cardiac disorders) | 1 (1)
RA lead noise (Cardiac disorders) | 1 (1)
RA lead oversensing or lead noise (Cardiac disorders) | 1 (1)
Twiddler's syndrome (Cardiac disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2010-11-16): https://cdn.clinicaltrials.gov/large-docs/64/NCT00810264/Prot_000.pdf
  • Statistical Analysis Plan (2019-04-26): https://cdn.clinicaltrials.gov/large-docs/64/NCT00810264/SAP_001.pdf